CLINICAL TRIAL: NCT05577234
Title: Contribution of Animal-assisted Intervention in Oral Healthcare for Disabled Patients
Brief Title: Contribution of Animal-assisted Intervention in Oral Healthcare for Disabled Patients (YODA)
Acronym: YODA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP220662; 2022-A00871-42 (Other: ID-RCB Number)
Record Dates: First submitted 2022-09-05; First posted 2022-10-13 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Autism
Keywords: Animal-assisted therapy; child; autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Animal-assisted intervention (Experimental): The dog accompanied by the zootherapist will participate in the care of the sessions. During these sessions, the dog will be brought into the child's presence in the waiting room until the end of the dental consultation.
  Interventions: Other: Animal-assisted intervention; Behavioral: Venham scale modified by Veerkamp
- Standard care (Other): The treatment sessions will only involve the use of conventional behavioural strategies.
  Interventions: Behavioral: Venham scale modified by Veerkamp

INTERVENTIONS:
Other: Animal-assisted intervention — The dog accompanied by the zootherapist will participate in the care of sessions 1 and 2. During these two sessions, the dog will be present with the child in the waiting room until the end of the dental consultation. Session 3 will take place without the dog being present.The usual management with conventional behavioural strategies and possible administration of MEOPA will be implemented during the 3 treatment sessions.
  Arms: Animal-assisted intervention
Behavioral: Venham scale modified by Veerkamp — The Venham scale modified by Veerkamp, based on observation of one's behaviour and used in current practice, ranges from 0 (relaxed) to 5 (totally disconnected from the reality of danger).

SUMMARY:
The purpose of this study is to determine whether animal-assisted therapy during 2 care sessions then facilitates conventional ambulatory management without animal assistance in anxious uncooperative children with autism.

DETAILED DESCRIPTION:
The particularity of some disabled patients, especially those with an autism spectrum disorder, is represented by anxiety, which can range from a slight tension to screaming or even extreme agitation. This behavior can make therapeutic management difficult, both for the patient and the caregiver. This is particularly true for oral health care, where the cooperation of the patient is essential. Conventional behavioral approaches, with implementation of a multitude of adaptive strategies, has a fundamental role to play. With disabled patients, these techniques are most often based on non-verbal or para-verbal communication rather than on linguistic procedures. In this context, an Animal Assisted Intervention could be of major help. The primary outcome is average child anxiety during the session assessed by the Venham scale modified by Veerkamp measured at the end of the third session of care (without animal-assisted therapy).

ELIGIBILITY:
Inclusion Criteria:

* Minors aged ≥ 6 to ≤ 17 years,
* Carriers of Autism Spectrum Disorder.
* Child with an average Venham scale score ≥ 3 at the end of the care of the inclusion session
* Who accept the presence of the dog
* Who declare having been in contact with a dog in the past
* Consent from the child's legal guardians for the child's participation in the study,
* Be affiliated to a social security scheme in their own name or be the legal guardian of a person with parental authority.
* A state of health requiring a simple, non-complex dental procedure (preventive, carious, traumatic or orthodontic care, excluding complex surgery in the operating theatre)
* A state of health requiring a dental treatment protocol consisting of at least 3 scheduled treatment sessions spaced at least 7 days and no more than 21 days apart.

Exclusion Criteria:

* Child with dog allergy
* Cynophobia
* Who claims never to have been exposed to a dog (allergy risk not assessed)
* Patient on AME

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2023-03-24 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
Average anxiety | through study completion, an average of 3 months
  Average anxiety of the child during the session assessed by the Venham scale modified by Veerkamp measured at the end of the third treatment session (without animal assisted intervention). Score on a scale : Min = 0 Max = 5 : 0 = relaxed, 1 = uneasy, 2 = tense, 3 = unwilling, 4 = very troubled, 5 = totally out of touch

SECONDARY OUTCOMES:
Evaluate the success of the care session (complete achievement of the planned objective) | at the end of each follow-up visit, on average 3 months
  Overall success of the session: dental care completed in its entirety
Validate the use of MEOPA administration | at the end of each follow-up visit, on average 3 months
  Use of MEOPA: administration of MEOPA during the session
Assess the types of acts for which animal assisted intervention reduces the child's anxiety | at the end of each follow-up visit, on average 3 months
  Types of procedures for which animal assisted intervention reduces anxiety: assessment of anxiety by the Venham scale modified by Verkamp measured at the end of each type of procedure : waiting room, entry into practice, X-rays, anaesthesia, placement of the dam, use of rotary instruments
Assessing the safety of animal assisted intervention for oral care | at the end of each follow-up visit, on average 3 months
  Occurrence of undesirable events associated with the animal assisted intervention, including infectious events of the zoonosis type (assessment by the practitioner at the beginning of each session and by the accompanying person who must report to the practitioner any manifestation that has appeared since the last session), episodes of agitation linked to the presence of the dog, bites.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc TRELUYER, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Bretonneau - Service d'odontologie, Paris, France

IPD SHARING:
Plan to Share IPD: No